CLINICAL TRIAL: NCT03956732
Title: Effects of Milk Protein and Vitamin D on Children's Growth and Health (D-pro)
Brief Title: Effects of Milk Protein and Vitamin D on Children's Growth and Health
Acronym: D-pro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: University of Aarhus (Other); Arla Foods (Industry); Arla Foods Ingredients (Unknown)
Responsible Party: Principal Investigator, Camilla Trab Damsgaard, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D224
Record Dates: First submitted 2019-05-16; First posted 2019-05-21 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Bone Health; Muscle Function; Cardiometabolic Health; Appetite Regulation
Keywords: Child Nutrition; Dietary recommendations; Milk protein; Vitamin D; Bone mineral density; Muscle strength; Immune defence
MeSH Terms: interventions — Milk Proteins; Vitamin D; Culture Media

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: D-pro will be double-blinded in respect to D vitamin supplementation or placebo, whereas the allocation of yoghurt with high versus medium milk protein content will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High protein yoghurt and vitamin D supplement (Experimental): Subjects will receive high protein yoghurt and vitamin D tablets.
  Interventions: Dietary Supplement: Milk Protein (high); Dietary Supplement: Vitamin D
- High protein yoghurt and placebo supplement (Experimental): Subjects will receive high protein yoghurt and placebo tablets of identical appearance and taste but without vitamin D.
  Interventions: Dietary Supplement: Milk Protein (high)
- Medium protein yoghurt and vitamin D supplement (Experimental): Subjects will receive medium protein yoghurt and vitamin D tablets.
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: Milk Protein (medium)
- Medium protein yoghurt and placebo supplement (Placebo Comparator): Subjects will receive medium protein yoghurt and placebo tablets of identical appearance and taste but without vitamin D.
  Interventions: Dietary Supplement: Milk Protein (medium)

INTERVENTIONS:
Dietary Supplement: Milk Protein (high) — High protein yoghurt which contains approx. 10 g protein per 100 g. Participants will be asked to consume 300 g (=3 dl) 6 days a week.
  Arms: High protein yoghurt and placebo supplement; High protein yoghurt and vitamin D supplement
Dietary Supplement: Vitamin D — One daily tablet containing 20 μg of vitamin D3, cholecalciferol.
  Arms: High protein yoghurt and vitamin D supplement; Medium protein yoghurt and vitamin D supplement
Dietary Supplement: Milk Protein (medium) — Ordinary yoghurt containing approx. 3.3 g protein per 100 g. Participants will be asked to consume 300 g (=3 dl) 6 days a week.
  Arms: Medium protein yoghurt and placebo supplement; Medium protein yoghurt and vitamin D supplement

SUMMARY:
The purpose of D-pro is to investigate the combined and separate effects of milk protein and vitamin D on bone health, growth, muscle function, body composition and cardiometabolic health in 6-8-year-old children.

DETAILED DESCRIPTION:
The D-pro study investigates the effects of high or medium intakes of milk protein, and vitamin D supplements or placebo, in healthy 6-8 year-old Danish children. The study is a 2×2-factorial randomized controlled trial with 4 study arms. The subjects will be randomly allocated to receive yoghurt products with either high or medium protein content (300g/day, 6 days/week) and to receive tablets with either vitamin D (20 μg/day) or placebo for 24 weeks. Measurements and biological sampling will be performed at baseline and at the end of the intervention.

The primary outcome will be bone mineral density (BMD). The investigators will also measure effects on children's muscle function, cardiometabolic health, body composition, growth and growth factors, nutrient status, immune defence and risk of acute respiratory tract infections, as well as appetite hormones. The investigators will also assess potential sex-specific effects and the potential modifying effect of genotype.

ELIGIBILITY:
Inclusion Criteria:

Children must:

* Be 6-8 years of age at the start of the intervention
* Be healthy
* Have a frequent intake of milk and yoghurt products, corresponding to at least ¼ liter a day
* Like yoghurt and high protein yoghurt ("skyr")
* Be of white, Danish or European origin

Moreover:

* The family must not be planning a winter vacation south of a latitude of 50° North
* The child must speak and understand Danish in order to understand the study procedures
* At least one parent must read, speak and write Danish

Exclusion Criteria:

* Known or suspected allergy or intolerance to milk or milk components
* Chronic illness or disease that may affect study outcomes
* Chronic intake of medicine that may affect study outcomes
* Use of vitamin D-containing supplements >3 days/week the 2 last months and use of any vitamin D-containing supplements the last 1 month before intervention start
* Concomitant participation in other studies involving dietary supplements or blood sampling
* Living in a household with another participating child

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density (BMD) | 24 weeks
  Measured by dual energy x-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Bone Mineral Content (BMC) | 24 weeks
  by DXA
Fat mass index | 24 weeks
  by DXA
Fat free mass index | 24 weeks
  by DXA
Bone area | 24 weeks
  by DXA
Height | 24 weeks
  by stadiometer
Waist circumference | 24 weeks
Insulin-like Growth Factor 1 (IGF-1) | 24 weeks
  by fasting blood sample
Insulin-like growth factor-binding protein 3 (IGFBP-3) | 24 weeks
  by fasting blood sample
Serum calcium | 24 weeks
  by fasting blood sample
Osteocalcin | 24 weeks
  by fasting blood sample
Parathyroid hormone (PTH) | 24 weeks
  by fasting blood sample
Bone-specific alkaline phosphatase | 24 weeks
  by fasting blood sample
C-terminal telopeptide of type 1 collagen in serum (s-CTX) | 24 weeks
  by fasting blood sample
Maximal leg press strength | 24 weeks
  Measured by isometric leg press
Maximal jumping height | 24 weeks
  Measured by squat jump with linear encoder
Maximal jumping length | 24 weeks
  Measured by standing long jump
Maximal grip strength | 24 weeks
  Measured by hand grip dynamometer
Muscle endurance | 24 weeks
  Measured by 30 sec. sit-to-stand
Blood pressure | 24 weeks
Hemoglobin A1c (HbA1c) | 24 weeks
  by fasting blood sample
Glucose | 24 weeks
  by fasting blood sample
Insulin | 24 weeks
  by fasting blood sample
Total cholesterol | 24 weeks
  by fasting blood sample
High density lipoprotein cholesterol (HDL cholesterol) | 24 weeks
  by fasting blood sample
Low density lipoprotein cholesterol (LDL cholesterol) | 24 weeks
  by fasting blood sample
Triacylglycerol (TG) | 24 weeks
  by fasting blood sample

OTHER OUTCOMES:
Physical activity | 24 weeks
  by accelerometry
C-peptide | 24 weeks
  by fasting blood sample
Vitamin D binding protein | 24 weeks
  by fasting blood sample
Serum 25(OH) vitamin D | 24 weeks
  by fasting blood sample
1,25(OH)2vitamin D | 24 weeks
  by fasting blood sample
Urea | 24 weeks
  by fasting blood sample
Interleukin-6 (IL-6) | 24 weeks
  by fasting blood sample
Interleukin-1β (IL-1β) | 24 weeks
  by fasting blood sample
Tumor necrosis factor a (TNF-a) | 24 weeks
  by fasting blood sample
Leptin | 24 weeks
  by fasting blood sample
Adiponectin | 24 weeks
  by fasting blood sample
High sensitivity C-reactive protein (hsCRP) | 24 weeks
  by fasting blood sample
Immune cell counts | 24 weeks
  by fasting blood sample
Immuno-active peptides in nasal fluid | 24 weeks
  by nasal fluid sample
Immuno-active peptides in blood | 24 weeks
  by fasting blood sample
Respiratory tract infections | 24 weeks
  by questionnaires
Dietary intake | 24 weeks
  By 4-day dietary record
Vitamin D and calcium intake | 24 weeks
  By food frequency questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Camilla T Damsgaard, Assoc Prof, Principal Investigator — University of Copenhagen; Christian Mølgaard, Prof, Study Chair — University of Copenhagen; Mette Hansen, Assoc Prof, Study Chair — Institute of Public Health, Aarhus University, Denmark
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Frederiksberg, Denmark

REFERENCES:
- [Derived] Clerico JW, Thams L, Stounbjerg NG, Hauger H, Damsgaard CT, Molgaard C. Effects of vitamin D supplementation on acute respiratory tract infections in 6-8-year-old children: a randomized clinical trial. Eur J Nutr. 2025 May 1;64(4):170. doi: 10.1007/s00394-025-03674-1. PMID 40310565
- [Derived] Thams L, Hvid LG, Stounbjerg NG, Brond JC, Molgaard C, Damsgaard CT, Hansen M. Vitamin D supplementation and increased dairy protein intake do not affect muscle strength or physical function in healthy 6-8-year-old children: the D-pro randomized trial. Eur J Nutr. 2022 Oct;61(7):3613-3623. doi: 10.1007/s00394-022-02912-0. Epub 2022 May 28. PMID 35643873
- [Derived] Thams L, Stounbjerg NG, Hvid LG, Molgaard C, Hansen M, Damsgaard CT. Effects of high dairy protein intake and vitamin D supplementation on body composition and cardiometabolic markers in 6-8-y-old children-the D-pro trial. Am J Clin Nutr. 2022 Apr 1;115(4):1080-1091. doi: 10.1093/ajcn/nqab424. PMID 35015806
- [Derived] Stounbjerg NG, Thams L, Hansen M, Larnkjaer A, Clerico JW, Cashman KD, Molgaard C, Damsgaard CT. Effects of vitamin D and high dairy protein intake on bone mineralization and linear growth in 6- to 8-year-old children: the D-pro randomized trial. Am J Clin Nutr. 2021 Dec 1;114(6):1971-1985. doi: 10.1093/ajcn/nqab286. PMID 34581765